CLINICAL TRIAL: NCT01000870
Title: An Exploratory, Open-label, Non-randomized Phase 0 Study to Evaluate Efficacy & Safety of MNI-513 Positron Emission Tomography for Detection/Exclusion of Cerebral Amyloid Beta in Patients w/ Alzheimer Disease Compared to Healthy Volunteers
Brief Title: Safety and Efficacy of Positron Emission Tomography Imaging With MNI-513
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Results did not show reason to continue with study
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Danna Jennings, MD / Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MNI-513-01
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Access MNI-513 and PET Imaging (Experimental)
  Interventions: Drug: MNI-513-01

INTERVENTIONS:
Drug: MNI-513-01 — Subjects will be administered a single IV injection of IMP with a total activity amounting to 300MBq (8.1 mCi) +/- 20% of MNI-513 followed by PET imaging.

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of MNI-513 positron emission tomography (PET) for detection/exclusion of cerebral amyloid beta in patients with Alzheimer's disease compared to healthy volunteers.

DETAILED DESCRIPTION:
To determine diagnostic efficacy of the MNI-513 PET scans in differentiating between patients with probable AD and HVs on the basis of neocortical tracer binding pattern, the PET scans will be visually assessed by a nuclear physician experienced in the field of neuro-imaging. PET scan findings will be classified either as abnormal (i.e., significant neocortical uptake in predefined regions) or as normal (i.e. no significant neocortical uptake in predefined regions). The nuclear physician will be unaware of the clinical diagnosis.

ELIGIBILITY:
INCLUSION CRITERIA: ALZHEIMER & HEALTHY VOLUNTEERS

1. is a man or woman and is ≥ 55 of age, whereby females must be without childbearing potential (confirmed by either: age ≥ 60; or history of surgical sterilization or of hysterectomy, or last spontaneous bleeding at least 2 years prior to the study start)
2. has at least 6 years of education
3. is able to provide informed consent or assent, and exhibits adequate visual, auditory and communication capabilities to enable compliance with study procedures. This includes performing the psychometric testing and being able to lie down flat in the PET scanner
4. possesses a general health that permits adequate compliance with all study procedures as ascertained by a detailed review of the medical history, laboratory and physical examination findings, which must be performed within 28 days prior to administration of IMP
5. the subject, or the subject and caregiver (for probable AD patients) will be compliant and have a high probability of completing the study in the opinion of the investigator
6. informed consent has been signed and dated (with time) by the subject and/or the subject's caregiver (for probable AD patients)

INCLUSION CRITERIA: HEALTHY VOLUNTEERS ONLY

1. has no evidence of cognitive impairment as indicated by a clinical dementia rating (CDR, [Hughes et al. 1993]) score of 0 (zero) and a score of ≥ 28 in the Mini-Mental Status Examination (MMSE, [Folstein et al. 1975])
2. has in the CERAD neuropsychological test battery [Welsh et al. 1994] a z- score of

   ≥ (-1.00) for each subtest (except for the MMSE which is covered by criterion 1 above)
3. has MRI brain scan that has been judged as "normal (age- appropriate)" including ARWMC scale [Wahlund et al. 2001] scores supporting the lack of cerebrovascular disease (e.g., a white matter lesion score of 0 or 1 or 2 and a basal ganglia score of 0 or 1) and a Scheltens scale [Scheltens et al. 1992] verifying the lack of cerebral atrophy (e.g. bilateral temporal lobe atrophy visual score of 0 or 1)

INCLUSION CRITERIA: PROBABLE ALZHEIMER DISEASE ONLY

1. presents with positive assessment for dementia of Alzheimer's type in accordance with the DSM-IV-TR and probable AD according to the NINCDS-ADRDA criteria and fulfils none of the exclusion criteria of either (see Appendix 1,2)
2. does not fulfill the ICC criteria for probable DLB (Appendix 3), the NINDS-AIREN for probable Vascular dementia (Appendix 5), or the Neary [Neary et al. 1998] criteria for FTD (Appendix 4)
3. has a CDR [Hughes et al. 1993] score of 0.5, 1 or 2
4. MRI brain scan findings that do not reveal changes indicative of stroke and/or generalized cerebrovascular disease (e.g., the ARWMC scale) changes limited to: a white matter lesion score of 0 or 1 or 2 and a basal ganglia score of 0 or 1)
5. has a caregiver who is willing and able to attend all study visits and perform the psychometric tests requiring the presence of a caregiver

EXCLUSION CRITERIA: ALZHEIMER DISEASE & HEALTHY VOLUNEERS

1. has any contraindication to MRI examination, e.g. metal implants or phobia as determined by the onsite radiologist performing the scan
2. is scheduled for surgery and/or another invasive procedure within the time period of up to 24 hours following IMP application
3. is allergic to the IMP or any of its constituents and/or has a history of severe allergic reactions to drugs or allergens (e.g. patients / volunteers with allergic asthma)
4. is critically ill and/or medically unstable and whose clinical course during the observation period is unpredictable, e.g. patients / volunteers within 14 days of myocardial infarction or stroke, unstable patients / volunteers with previous surgery (within 7 days), patients with advanced heart insufficiency (NYHA stage IV), or with acute renal failure
5. has a history of exposure to any radiation >15 mSv/year (e.g. occupational or radiation therapy)
6. is receiving drug therapy or other treatment that is known to lead to greatly fluctuating values of the hematological or chemical laboratory parameters or to severe side effects (e.g. chemotherapy)
7. has received anti-amyloid drug therapy.
8. has received any contrast material (X-ray, MRI) or radiopharmaceuticals within 48 hours prior to the application of the IMP or for whom application of such a substance is planned for the 24 hours following IMP administration
9. has been previously enrolled in this study or participated in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening, and/or any radiopharmaceutical within 10 radioactive half-lives prior to IMP administration
10. has a brain tumor or other intracranial lesion, a disturbance of CSF circulation (e.g., normal pressure hydrocephalus) and/or a history of head trauma or brain surgery
11. has an inflammatory or infectious CNS disease, e.g. multiple sclerosis, HIV, syphilis, or Creutzfeld-Jacob disease
12. has a history, physical, laboratory or imaging findings indicative of a significant neurological or psychiatric illness (for patients - other than AD)
13. has another disease that can cause disturbance of brain function (e.g. vitamin B12 or folic acid deficiency, disturbed thyroid function)
14. has a history of alcohol or drug abuse 15 has history of severe persistent depression

16.clinically significant hematologic indices that may put subject at increased risk for bleeding

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of MNI-513 positron emission tomography (PET) for detection/exclusion of cerebral amyloid beta in patients with Alzheimer's disease compared to healthy volunteers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States